CLINICAL TRIAL: NCT04235023
Title: PTP1B Implication in the Vascular Dysfunction Associated With Obstructive Sleep Apnea
Acronym: MacroSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC19-0226
Record Dates: First submitted 2020-01-07; First posted 2020-01-21 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Sleep Apnea; Inflammation; Atherosclerosis
Keywords: PTP1B; macrophage
MeSH Terms: conditions — Sleep Apnea Syndromes; Inflammation; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: patients with OSA 'apnea hypopnea index ≥ 15 per hour) as compared to controls (an apnea hypopnea index < 15 per hour)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSA patients (Other): 30 patients investigated for suspected OSA with an apnea hypopnea index ≥ 15 per hour
  Interventions: Other: myeloid PTP1B expression analysis
- non OSA patients (Other): 30 patients investigated for suspected OSA with an apnea hypopnea index < 15 per hour
  Interventions: Other: myeloid PTP1B expression analysis

INTERVENTIONS:
Other: myeloid PTP1B expression analysis — peripheral blood macrophage PTP1B expression

SUMMARY:
Obstructive sleep apnea (OSA) syndrome is associated with increased vascular dysfunction and atherosclerosis. Especially, it has been shown that OSA associated intermittent hypoxia represents a pro inflammatory stimulus resulting in macrophage polarization.

Protein tyrosine phosphatase 1B (PTP1B) is a negative regulator of insulin signaling pathways involved in atherosclerosis. It has been shown that myeloid PTP1B deficiency protects against atherosclerosis.

As hypoxia has also been shown to increase PTP1B expression and activity, this study will evaluate the myeloid PTP1B expression and activity in patients with OSA as compared to controls and will investigate myeloid PTP1B involvement in the vascular pro inflammatory precess described in OSA.

ELIGIBILITY:
Inclusion Criteria:

* Overnight polysomnographic recording for suspected OSA
* Apnea hypopnea index ≥ 15 per hour for OSA patients
* Apnea hypopnea index < 15 per hour for non OSA patients

Exclusion Criteria:

* past history of cardiovascular diseases
* diabetes
* dyslipidemia
* hypertension
* obesity (body mass index > 35 kg/m2
* past history or ongoing inflammatory diseases
* cognition impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
myeloid PTP1B expression | baseline
  Peripheral blood will be collected from OSA and non OSA patients. Macrophage will be isolated by specific centrifugation. PTP1B expression will be assessed by Western Blot.
myeloid PTP1B activity | baseline
  Peripheral blood will be collected from OSA and non OSA patients. Macrophage will be isolated by specific centrifugation. PTP1B activity will be assessed by specific colorimetric assay.

SECONDARY OUTCOMES:
PTP1B exosomal expression. | baseline
  Peripheral blood will be collected from OSA and non OSA patients. Exosomes will be isolated by consecutive centrifugations. PTP1B expression will be assessed by Western Blot.
in vitro PTP1B implication on macrophage inflammatory response | baseline
  Macrophage isolated from patients will be stimulated by pro inflammatory agents (IL6, TNF alpha) in the presence and absence of PTP1B inhibitor (MSI-1436). The inflammatory response will be assessed by measuring inflammatory cytokines in the supernatant by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Trzepizur, MD Ph D, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided